CLINICAL TRIAL: NCT00722228
Title: Autologous and Allogeneic Whole Cell Cancer Vaccine for Metastatic Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0359-08-HMO-CTIL
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Ovarian Cancer; Gastric Cancer; Breast Cancer; Lung Cancer; Kidney Cancer; Melanoma
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Breast Neoplasms; Lung Neoplasms; Kidney Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous or Allogeneic tumor cells (Experimental): Intervention: 5 vaccine doses, 3 weeks apart, injected subcutaneously.
  Interventions: Biological: Autologous or Allogeneic tumor cells

INTERVENTIONS:
Biological: Autologous or Allogeneic tumor cells — Five vaccine doses, injected subcutaneously at 3-week intervals. Each dose is composed of irradiated and DNP-conjugated tumor cells.

SUMMARY:
This study is based on the finding that tumor cells that are grown in the laboratory can be modified in such a way that, when injected to the patient, they will stimulate his/her immune response. This approach will be evaluated in patients with melanoma and colorectal, gastric, ovarian, breast, lung and kidney epithelial cancer. Tumor cells grown in the laboratory will be modified to make them stimulatory to the immune system, irradiated to kill them, and injected to the patient eight times at two-week intervals. This protocol is expected to prolong survival of metastatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* One of the following metastatic cancers: Melanoma, breast, ovary, colorectal, gastric, lung or kidney
* Above 18 years of age
* Failure of at least one chemotherapy protocol
* Clinical performance status of ECOG 0,1
* Absolute neutrophil count greater than 1000/mm3
* Serum ALT/AST less than three times the upper limit of normal
* Serum creatinine less than or equal to 1.6 mg/dl.
* Must be able to understand and sign the Informed Consent document

Exclusion Criteria:

* Below 18 years of age
* Women who are pregnant
* Life expectancy of less than three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-07 (Actual); Primary Completion 2025-03 (Actual); Study Completion 2027-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel